CLINICAL TRIAL: NCT02345369
Title: Does Static Locking of Set Screws in Intramedullary Fixation of Intertrochanteric Fractures Prevent Shortening of Intertrochanteric Hip Fractures?
Brief Title: Locked Versus Unlocked Set Screws in Intramedullary Fixation of Intertrochanteric Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change in surgical implant use, loss of subinvestigator
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Jennifer Victory, RN, CCRC, Clinical Research Nurse Supervisor, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1095
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Locked Set Screw (Active Comparator): In this arm, subjects who have sustained an intertrochanteric hip fracture (OTA classification A2 and A3) will undergo fixation with an intramedullary hip screw with locking of the set screw.
  Interventions: Device: Locked Set Screw
- Unlocked Set Screw (Active Comparator): In this arm, subjects who have sustained an intertrochanteric hip fracture (OTA classification A2 and A3) will undergo fixation with an intramedullary hip screw without locking of the set screw.
  Interventions: Device: Unlocked Set Screw

INTERVENTIONS:
Device: Locked Set Screw — Fixation of hip fracture with intramedullary hip screw with locking of the set screw
  Arms: Locked Set Screw
Device: Unlocked Set Screw — Fixation of hip fracture with intramedullary hip screw without locking of the set screw
  Arms: Unlocked Set Screw

SUMMARY:
The purpose of this study is to look at the effect of locking or not locking a set screw when placing a rod and screws device in the thigh bone and hip to fix hip fractures. The set screw is an extra screw in the device that will not allow the screw that goes into the ball of the ball and socket joint in the hip to slide at all in relation to the rod in the thigh bone, which it goes through. It is not known whether it is better to lock the set screw (not allow sliding of the hip screw) or leave it unlocked (allow sliding of the hip screw). Participants in this study are patients with intertrochanteric hip fractures receiving standard care for this injury (lining the fracture up in a normal position and inserting a rod in the thigh bone with a screw that goes through the rod into the ball of the ball and socket of the hip). Patients who consent to participate will be randomized to one of two arms : 1. Set screw is unlocked or 2. Set screw is locked. Participants will all get standard postoperative care and standard postoperative xrays.

DETAILED DESCRIPTION:
Intramedullary hip screw devices can be inserted with and without locking of the set screw, with the purpose of the set screw to minimize shortening of the femoral neck by rigidly positioning the head screw that inserts into the femoral head. Rigid locking of the lag screw may also limit the ability of the fracture fragments to compress against each other gradually with weight bearing and this potentially could reduce healing at the fracture site. Alternatively, more settling at the fracture site may allow more reliable healing while allowing more shortening of the femoral neck at the fracture site. Shortening of the femoral neck fracture can result in gait disturbances and poor hip function, while delay in healing can contribute to hardware failure and need for revision surgery. The benefit of placing the set screw in intramedullary hip screw fixation has not been clearly established in the literature. To date, there has been no study addressing this question, and the decision to lock, or not lock the screw is based on individual surgeon discretion. This study will help to clarify this decision point in the treatment of intertrochanteric hip fractures with the Intertan (Smith and Nephew, Memphis, Tn) intramedullary nail. This will lead to better patient outcomes, and help clarify the standard of care in these very common fracture patterns.

Subjects who have sustained an intertrochanteric hip fracture (OTA classification A2 and A3) will be randomized to undergo fixation with an intramedullary hip screw with and without locking of the set screw. These subjects will be blinded to the study group and will be treated as per standard of care after fixation of a hip fracture with xrays immediately after surgery, at 1-2 weeks, 6 weeks, and then 3 and 6 months post operatively. As per standard care additional xrays would be indicated until union of the fracture if there is delayed healing. Femoral neck shortening will be measured radiographically with femoral neck offset and the femoral neck shaft angle to be measured radiographically based on standardized computerized measurements from the xray images. TraumaCad software (Voyanthealth, Westchester, Il) will be utilized to obtain standardized measurements. A blinded subinvestigator will review the participants' x-rays and make the measurements required to determine the study outcomes. Time to radiographic union and any occurrence of hardware failure, nonunion and malunion will be noted. Demographic data including age, gender, smoking history, and medical comorbidities will be collected based on chart review. Subjective outcome scores (modified Harris hip score) will be collected at 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

All subjects 18 years or older who are:

* mentally competent to give consent and complete the follow up questionnaires
* being treated for an intertrochanteric hip fracture,
* classified as Arbeitsgemeinschaft für Osteosynthesefragen/Orthopaedic Trauma Association (AO/OTA) 31-A2 or A3
* plan to be treated with an intramedullary hip screw

Exclusion Criteria:

* infection in the involved joint or surrounding soft tissues,
* pathological fractures as a result of metastatic or primary bone tumors, progressive or debilitating neurological conditions resulting in significant movement or gait disorders, congenital bone disorders or heritable bone disorders (excluding osteoporosis and osteopenia),
* severe dementia,
* nonambulatory patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: jocelyn wittstein, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment ended when lead surgeon left the institution & types of implants used by institution were changed
Period: Overall Study
Arm/Group | Locked Set Screw | Unlocked Set Screw
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: study terminated when lead surgeon left institution
Groups:
- Total: Total of all reporting groups
Arm/Group | Locked Set Screw | Unlocked Set Screw | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Femoral Neck Shortening
Description: Femoral neck shortening will be measured radiographically with femoral neck offset and the femoral neck shaft angle to be measured radiographically based on standardized computerized measurements based off of PACs images. TraumaCad software (Voyanthealth, Westchester, Il) will be utilized to obtain standardized measurements.
Time Frame: 6 months
Population: no outcomes to report
Arm/Group | Locked Set Screw | Unlocked Set Screw
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Radiographic Union
Description: Time to radiographic union and any occurrence of hardware failure, nonunion and malunion will be noted
Time Frame: 6 months
Population: no outcomes to report
Arm/Group | Locked Set Screw | Unlocked Set Screw
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Harris Hip Score
Description: Subjective outcome scores (modified Harris hip score) will be collected at 3 and 6 months after surgery.
Time Frame: 6 months
Population: no outcomes to report
Arm/Group | Locked Set Screw | Unlocked Set Screw
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: NA - study terminated
Description: NA - study terminated
Arm/Group | Locked Set Screw | Unlocked Set Screw
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes